CLINICAL TRIAL: NCT00985881
Title: Mechanically-induced Stochastic Resonance to Improve Amputee Gait
Brief Title: Use of Subtle Vibration to Improve Walking Ability by Lower Limb Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: A4376-R
Record Dates: First submitted 2008-03-25; First posted 2009-09-29 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Amputation; Diabetes Complications
Keywords: Artificial limbs; Gait; Posture; Prosthesis; Vibration
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: stochastic resonance (Experimental): Mechanical stochastic resonance
  Interventions: Device: Custom prosthetic socket with mechanical vibrators (stochastic resonance)
- Arm 2: current clinical practice (Other): Current clinical practice
  Interventions: Device: Conventional prosthetic socket (current clinical practice)

INTERVENTIONS:
Device: Custom prosthetic socket with mechanical vibrators (stochastic resonance) — Application of mechanically-induced sub-threshold vibration applied to the amputee's residual limb using a custom prosthetic limb system
  Arms: Arm 1: stochastic resonance
Device: Conventional prosthetic socket (current clinical practice) — No sub-threshold vibration applied to residual limb. Amputee wears conventional prosthetic socket.
  Arms: Arm 2: current clinical practice

SUMMARY:
The purpose of this study is to determine if subthreshold vibration, when applied to the residual limb of a lower limb amputee through their prosthetic socket, can sufficiently enhance peripheral sensation to result in an improved ability to balance and walk.

DETAILED DESCRIPTION:
One of the many complications of diabetes is the loss of sensation in the feet. This sensory deficit can negatively impact the postural stability and mobility of non-amputees, since without feedback, it is simply more difficult to stand and walk. For lower limb amputees, the problem is compounded. These patients often have difficulty with prosthetic limb placement during maneuvering tasks, exhibit dramatic increases in the movement of their center of pressure during quiet standing, and both clinical and observational gait analysis reveal significant changes in their gait pattern relative to non-amputees.

The investigators' work proposes to explore the use of a novel prosthetic intervention for diabetic lower limb amputees. The investigators hypothesize that the intervention will sufficiently enhance proprioception to result in measurably improved postural stability and locomotor function for these patients. The intervention is based on a phenomenon known as stochastic resonance, whereby the application of sub-threshold vibration enables mechano-receptors previously unable to respond to stimuli to become more susceptible to depolarization. For Veterans with neuropathic proprioceptive losses, stochastic resonance may facilitate a functional response from subtle stimuli where gross inputs were formerly required.

ELIGIBILITY:
Inclusion Criteria:

Amputee subjects:

* unilateral transtibial amputee of diabetic etiology,
* have been fit with a prosthesis and have used a prosthesis for at least one year,
* wear the prosthesis at least 4 hours per day,
* ambulate without upper extremity aids,
* have no history of injurious falls within the previous six months, and
* touch sensation measured by a 10 gauge Semmes-Weinstein Monofilament in the dermatomes of their residual limb.

Exclusion Criteria:

Subjects will be excluded if:

* they have a significant lower extremity pain condition, musculoskeletal disorder, or neurological deficit that interferes with their ability to pursue typical daily activities or alters their gait characteristics,
* their residual limb is ulcerated, or
* are currently using anticonvulsant medications for the treatment of neuropathic pain.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Gait variability | Testing with and without stochastic resonance will occur within a single laboratory visit on one day
  Self-selected walking speed (mean and standard deviation) in meters/second

CONTACTS AND LOCATIONS:
Overall Officials: Glenn K Klute, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study: Mechanically-induced Stochastic Resonance to Improve Amputee Gait — http://www.amputation.research.va.gov/